CLINICAL TRIAL: NCT06565377
Title: The Added Value of Multimodal Biopsychosocial Teleprehabilitation in People Undergoing Total Knee Arthroplasty: a Pilot/Feasibility Trial
Brief Title: Multimodal Biopsychosocial Teleprehabilitation for Total Knee Arthroplasty
Acronym: MULTIPREP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Vrije Universiteit Brussel (Other); Ziekenhuis Geel (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 12AV224N
Record Dates: First submitted 2024-08-05; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-07

CONDITIONS: Total Knee Arthroplasty
Keywords: total knee arthroplasty; knee replacement; prehabilitation
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal biopsychosocial teleprehabilitation (BPS-teleprehab) (Experimental): see intervention description
  Interventions: Behavioral: Multimodal biopsychosocial teleprehabilitation
- Best-evidence prehabilitation advice (control) (Active Comparator): see intervention description
  Interventions: Other: Best-evidence prehabilitation advice

INTERVENTIONS:
Behavioral: Multimodal biopsychosocial teleprehabilitation — Multimodal biopsychosocial teleprehabilitation containing (pain science and lifestyle) education, stress management and physical activity promotion, guided by shared decision making, motivational interviewing and solution focused therapy principles.
  Format: 4 preoperative and 1 postoperative one-on-one (tele-)conferencing sessions with a physical therapist, supplemented by an informational booklet.
  Other Names: prehabilitation
  Arms: Multimodal biopsychosocial teleprehabilitation (BPS-teleprehab)
Other: Best-evidence prehabilitation advice — Best-evidence prehabilitation advice in accordance with the NICE guideline on Joint Replacement (Primary): hip, knee and shoulder (2020), by means of an informational booklet.
  Arms: Best-evidence prehabilitation advice (control)

SUMMARY:
Knee replacement surgeries are one of the most frequently performed elective surgeries, with approximately 29,000 such procedures carried out annually in Belgium. Although these surgeries have been increasingly refined over the years, leading to better surgical outcomes, there is still room for improvement in terms of pre-surgical biopsychosocial patient preparation. Such preparation aims to optimally inform patients before their surgery and to start preparing them for rehabilitation and resumption of activities after surgery. Therefore, we aim to assess the added value and feasibility of prehabilitation within the knee replacement care pathway.

The primary objective is to investigate the feasibility, acceptability and safety of multimodal biopsychosocial teleprehabilitation (BPS-teleprehab) for people undergoing total knee arthroplasty (TKA).

The secondary objective is to explore the effect of BPS-teleprehab versus best-evidence preoperative advice for people undergoing TKA on activity outcomes, functioning, pain, symptoms of central sensitization, quality of life, cognitive-emotional factors, joint awareness, satisfaction with the surgery, healthcare and medication use and productivity loss.

The tertiary objective is to explore baseline associations between the collected outcome measures, demographics and medical data in people scheduled for TKA.

Furthermore, this pilot trial will inform potential protocol modifications in prepara- tion of an eventual fully powered randomized controlled trial to investigate the ef- fectiveness of BPS-teleprehab in people undergoing TKA.

ELIGIBILITY:
Inclusion Criteria:

* People scheduled for elective primary TKA at one of the participating hospitals;
* Being over 18 years old;
* Dutch speaking/reading

Exclusion Criteria:

* Doing activities that make them feel out of breath for 300 minutes or more per week on average;
* Orthopedic, neurological, cardiovascular or any other condition/comorbidity that leads to an overall contraindication for moderate physical activity;
* Cognitive impairment (≥11 on 6-item Cognitive Impairment Test and/or unable to understand the study instructions);
* Presence of uncontrolled inflammatory arthritides (e.g., rheumatoid arthritis, gout);
* Uncontrolled psychiatric disorders;
* Active cancer and/or active cancer treatment ((hormonal) maintenance therapy is allowed);
* People undergoing emergency (non-elective) TKA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Participation rate | assessed throughout the duration of the participant recruitment for the trial
  This will be calculated as the ratio of the number of patients participating in the study to the number of patients eligible for study participation.
Patient satisfaction with the intervention (feeling of contentment with the intervention) | at 6 weeks post-surgery
  This will be assessed by qualitative in-depth interviews with the study participants.
Incidence of treatment-emergent adverse events (safety and tolerability) | At the end of each intervention session + throughout the duration of the study
  After each intervention session, patients of the experimental group will be asked whether they experienced any side effects or unexpected events associated with the intervention. Furthermore, participants are encouraged to report any side effects/unexpected events to the study team at any time throughout the study.
Compliance with the one-on-one BPS-teleprehab sessions | Within one week after intervention completion
  The compliance rate for the teleprehabilitation sessions will be calculated as the ratio of the number of followed treatment sessions versus the number of planned treatment sessions.
Compliance with home exercises | Within one week after intervention completion
  Patients will be asked to log their home exercise sessions in an intervention log book. The compliance with these home exercise sessions is calculated as the ratio between the number of sessions performed and the number of sessions prescribed.
Feasibility of BPS-teleprehab in the clinical setting | through study completion
  The feasibility of BPS-teleprehab in the clinical setting will be investigated by qualitative focus group discussions with healthcare providers involved in the care trajectory of people undergoing total knee arthroplasty.

SECONDARY OUTCOMES:
Physical activity (objective measure) | Baseline, post-intervention (day 4-7 post-surgery), 6 weeks post-surgery, 6 months post-surgery (primary endpoint), 12 months post-surgery. Actigraphy data will be registered for 1 week prior to the assessment moment for the remaining outcomes.
  Actigraphy (Fitbit)
Physical activity (patient-reported outcome) | Baseline, post-intervention (day 4-7 post-surgery), 6 weeks post-surgery, 6 months post-surgery (primary endpoint), 12 months post-surgery. Actigraphy data will be registered for 1 week prior to the assessment moment for the remaining outcomes.
  International Physical Activity Questionnaire
Knee-specific pain and functioning | Baseline, post-intervention (day 4-7 post-surgery), 6 weeks post-surgery, 6 months post-surgery (primary endpoint), 12 months post-surgery.
  Knee Injury and Osteoarthritis Outcome Score (KOOS), scale from 0-100, higher scores indicate better outcome
Health-related quality of life | Baseline, 6 weeks post-surgery, 6 months post-surgery (primary endpoint), 12 months post-surgery.
  EQ-5D-5L (Euroqol); scale from 0-100; higher scores indicate better quality of life
Symptoms of central sensitization | Baseline, 6 months, 12 months post-surgery.
  Central Sensitization Inventory; scale from 0-100; higher scores indicate more symptoms of central sensitization
Pain catastrophizing | Baseline, post-intervention (day 4-7 post-surgery), 6 weeks post-surgery, 6 months post-surgery (primary endpoint), 12 months post-surgery.
  Pain Catastrophizing Scale; scale from 0-52; higher scores indicate higher levels of pain catastrophizing
Fear of movement and/or (re)injury | Baseline, post-intervention (day 4-7 post-surgery), 6 weeks post-surgery, 6 months post-surgery (primary endpoint), 12 months post-surgery.
  Tampa Scale for Kinesiophobia; scores from 17-68; higher scores indicate higher levels of fear of movement
Perceived Self-efficacy to exercise | Baseline, post-intervention (day 4-7 post-surgery), 6 weeks post-surgery, 6 months post-surgery (primary endpoint), 12 months post-surgery.
  Patient-reported questionnaire based on Neupert et al. (2009); scores from 9-36; higher scores indicate greater exercise-related self-efficacy
Joint awareness of the replaced joint | Post-intervention (day 4-7 post-surgery), 6 weeks post-surgery, 6 months post-surgery (primary endpoint), 12 months post-surgery.
  Forgotten Joint Score; sores from 0 to 100; high values translating to the patient successfully "forgetting" about their joint during activities of daily living
Satisfaction with surgery | Post-intervention (day 4-7 post-surgery), 6 weeks post-surgery, 6 months post-surgery (primary endpoint), 12 months post-surgery.
  4-item satisfaction questionnaire; scores from 0-20; higher scores indicating higher levels of contentment with the surgery
Total knee arthroplasty expectations | Baseline, post-intervention (day 4-7 post-surgery), 6 weeks post-surgery.
  Knee Replacement Expectations Survey; scores from 0-100; higher scores indicate higher expectations
Overall change following knee replacement surgery | Post-intervention (day 4-7 post-surgery), 6 weeks post-surgery, 6 months post-surgery (primary endpoint), 12 months post-surgery.
  Global Rating of Change; scores from -3 to +3; more positive scores indicate a more positive change
Healthcare and medication use | Baseline, 6 weeks post-surgery, 6 months post-surgery (primary endpoint), 12 months post-surgery.
  (Modified) Medical Consumption Questionnaire
Productivity loss/return to work | 6 months and 12 months post-surgery.
  Productivity Cost Questionnaire

OTHER OUTCOMES:
Focus groups with healthcare providers | Throughout the duration of the study
  Focus group discussions with healthcare providers involved in the care trajectory of people undergoing total knee arthroplasty concerning the feasibility of multimodal biopsychosocial teleprehabilitation in clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Huysmans, PhD, Principal Investigator — Vrije Universiteit Brussel
Locations (2):
- Belgium (2):
  - Ziekenhuis Geel, Geel, Antwerpen
  - Universitair Ziekenhuis Brussel, Brussels, Brussels Capital

IPD SHARING:
Plan to Share IPD: Yes
Open access data sharing is not possible due to the high degree of confidentiality of the pseudonymized medical and personal data. Data sharing (of pseudonymized data) is only permitted if all involved parties agree and if a data sharing agreement is signed. The research data need to be archived under restricted access due to the level of confidentiality of coded medical data. Requests for data sharing will be considered by the steering board. The informed consent allows for pseudonimyzed data sharing under these restricted conditions.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Requests for data sharing can be considered once the main results of the trial have been published.
Access Criteria: Requests for data sharing will be considered by the steering board of the study who will screen the applicants and (relevance of the) proposed research questions. If considered appropriate and relevant, a data sharing agreement will be composed in cooperation with our data protection officer and legal department.